CLINICAL TRIAL: NCT07363330
Title: Utidelone Combined With Toripalimab in Patients With Pretreated Recurrent or Metastatic Cervical Cancers: a Single-Arm, Phase II Study
Brief Title: A Phase II Study of Utidelone With Toripalimab in Advanced Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Hui Qiu, Head of Department, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025LCYJZX-ZD005
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer; Recurrent; Metastatic
Keywords: cervical cancer; recurrent / metastatic; Utidelone; Toripalimab; phase Ⅱ trial
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence; Neoplasm Metastasis | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Utidelone plus Toripalimab (Experimental): 1. Drug: Utidelone (1)Dosage: 30 mg/m² (2)Route of Administration: Intravenous drip (IV infusion) (3)Schedule: Administered once daily on Days 1-5 of each cycle. (4)Cycle Duration: 21 days (q3w).
  2. Drug: Toripalimab (1)Dosage: 240 mg (2)Route of Administration: Intravenous drip (IV infusion) (3)Schedule: Administered on Day 6 of each cycle. (4)Cycle Duration: 21 days (q3w).
  Interventions: Drug: Utidelone plus Toripalimab

INTERVENTIONS:
Drug: Utidelone plus Toripalimab — 1. Drug: Utidelone (1)Dosage: 30 mg/m² (2)Route of Administration: Intravenous drip (IV infusion) (3)Schedule: Administered once daily on Days 1-5 of each cycle. (4)Cycle Duration: 21 days (q3w).
  2. Drug: Toripalimab (1)Dosage: 240 mg (2)Route of Administration: Intravenous drip (IV infusion) (3)Schedule: Administered on Day 6 of each cycle. (4)Cycle Duration: 21 days (q3w).

SUMMARY:
This is a Phase II clinical trial to evaluate the safety and efficacy of Utidelone, a genetically engineered epothilone derivative, combined with Toripalimab, a PD-1 inhibitor, in patients with recurrent or metastatic cervical cancer who have progressed after standard treatments. The study will also assess the safety profile of this combination therapy. The primary objectives of this study include: (1) to determine the objective response rate (ORR), meaning whether the treatment can reduce the size of tumors or make them disappear, according to the RECIST 1.1 criteria; (2) to evaluate the safety of the treatment and document the side effects experienced by participants. This study is for individuals who: (1) are between 18 and 75 years old; (2) have a confirmed diagnosis of recurrent or metastatic cervical cancer; (3) have previously received at least one standard chemotherapy regimen that is no longer controlling the cancer; (4) are in generally good health, as determined by the study investigators. In this single-arm study, all participants will receive the same treatment: Utidelone will be administered by intravenous (IV) infusion over 1.5 hours, once a day for 5 consecutive days, in each 21-day treatment cycle; Toripalimab will be administered by IV infusion over 1.5 hours, once on Day 6 of each 21-day cycle. Participants may continue receiving the study drugs as long as they are benefiting from the treatment and side effects are manageable. Doctors will assess tumor size using imaging scans (like CT or MRI) every 6 weeks to monitor how the cancer responds to treatment. The study will take place at Zhongnan Hospital of Wuhan University and plans to include approximately 32 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent: Patients must voluntarily sign an informed consent form prior to any study-related procedures.
2. Age: Aged ≥18 years and ≤75 years.
3. Diagnosis: Histologically or cytologically confirmed recurrent or metastatic cervical carcinoma.
4. Performance Status: With an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Measurable Disease: With at least one measurable lesion as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
6. Prior Therapy:

   * Patients must have received at least one line of standard systemic chemotherapy for recurrent/metastatic disease, OR
   * Patients with rapid disease progression (occurring within 6 months) during or after prior neoadjuvant or concurrent chemoradiotherapy.
7. Treatment-Related Toxicity: Recovery from all toxicities related to prior anti-cancer therapies to ≤ Grade 1 (according to CTCAE v5.0). Patients with alopecia of any grade are eligible.
8. Adequate Hematological Function (within 1 week prior to enrollment, per local laboratory reference ranges):

   * White blood cell count (WBC) ≥ 2.5 × 10⁹/L.
   * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L.
   * Platelet count (PLT) ≥ 100 × 10⁹/L.
   * Hemoglobin (Hb) ≥ 9.0 g/dL (transfusion or erythropoietin use is permitted to meet this criterion).
9. Adequate Liver and Kidney Functions (within 1 week prior to enrollment, per local laboratory reference ranges):

   * Total bilirubin (TBIL) ≤ 1.5 × the upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN for patients with liver metastases).
   * Calculated creatinine clearance (Ccr) ≥ 60 mL/min.
10. Contraception: Patients of childbearing potential must agree to use highly effective contraception during the study and for at least 90 days after the last dose of study treatment. A negative serum or urine pregnancy test is required for female patients of childbearing potential within 7 days prior to enrollment.
11. Life Expectancy: Anticipated life expectancy of at least 12 weeks.
12. Compliance: Patients must be able and willing to comply with the study protocol for treatment and follow-up.

Exclusion Criteria:

1. Concurrent Malignancy: History of other active malignancies within the past 5 years, except for adequately treated basal cell carcinoma of the skin.
2. Recent Anti-cancer Therapy: Any anti-cancer therapy (including chemotherapy, radical radiotherapy, hormonal therapy, biological therapy, or anti-cancer Chinese herbal medicine) within 4 weeks prior to the initiation of study treatment.
3. Recent Major Surgery/Trauma: Major surgical procedure (excluding diagnostic biopsy) or significant traumatic injury within 4 weeks prior to the first dose of study drug, or anticipation of the need for major surgery during the study period.
4. Prior Neurotoxicity: History of ≥ Grade 3 neurological adverse reactions attributed to prior anti-microtubule therapy.
5. Symptomatic CNS Metastases: Patients with symptomatic central nervous system (CNS) metastases.
6. Pregnancy/Lactation: Women who are pregnant or breastfeeding.
7. Hypersensitivity: Known or suspected hypersensitivity to any component of the study drugs or their excipients.
8. Severe Comorbidities: Any uncontrolled or severe concurrent medical condition that, in the investigator's judgment, would preclude participation, including but not limited to:

   * Severe cardiovascular or cerebrovascular disease.
   * Uncontrolled diabetes mellitus or hypertension.
   * Active severe infection.
   * Active peptic ulcer disease.
   * Uncontrolled psychiatric illness/disorder.
9. General Exclusion: Any other condition or circumstance that, in the opinion of the investigator, would compromise the patient's safety or compliance, or make the patient unsuitable for study participation.
10. Contraindication to Steroids: Conditions for which corticosteroid use is contraindicated.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Tumor assessments are performed at baseline and every 6 weeks (± 3 days) until progression or start of new therapy. ORR is analyzed after all patients have completed at least 18 weeks of follow-up or experienced a study endpoint event.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of enrollment until first documented disease progression (per RECIST 1.1) or death from any cause, whichever occurs first, assessed up to approximately 24 months.
Time to Response (TTR) | From the date of enrollment to the first documented objective response (Complete or Partial Response per RECIST 1.1), assessed up to approximately 24 months.
Duration of Response (DoR) | From the date of first documented objective response (CR or PR) until documented disease progression or death due to underlying cervical cancer, assessed up to approximately 36 months.
Overall Survival (OS) | From the date of enrollment until death from any cause, assessed up to approximately 36 months.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From the first dose of study drug until 30 days after the last dose, assessed throughout the treatment period (up to approximately 24 months).
Incidence of Serious Adverse Events (SAEs) | From the first dose of study drug until 90 days after the last dose, assessed throughout the treatment and extended safety follow-up period (up to approximately 27 months).
Number of Participants With Clinically Significant Laboratory Abnormalities | Laboratory parameters are monitored at each 21-day treatment cycle from first dose until 30 days after the last dose (up to approximately 24 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qiao G, Liu Z, Ding H, Lu H, Lin F, Shi Y, Zheng L, Wang M, Chen Y, Deng Z, Yu L, Zhang Y, Yuan Y, Lin H, Ma L, Zhang J. Utidelone-based therapy in advanced or metastatic solid tumors after failure of standard therapies: a prospective, multicenter, single-arm trial. Am J Cancer Res. 2024 Sep 15;14(9):4514-4522. doi: 10.62347/OLES9793. eCollection 2024. PMID 39417192
- [Background] Xu B, Sun T, Zhang Q, Zhang P, Yuan Z, Jiang Z, Wang X, Cui S, Teng Y, Hu XC, Yang J, Pan H, Tong Z, Li H, Yao Q, Wang Y, Yin Y, Sun P, Zheng H, Cheng J, Lu J, Zhang B, Geng C, Liu J, Shen K, Yu S, Li H, Tang L, Qiu R; study group of BG01-1323L. Efficacy of utidelone plus capecitabine versus capecitabine for heavily pretreated, anthracycline- and taxane-refractory metastatic breast cancer: final analysis of overall survival in a phase III randomised controlled trial. Ann Oncol. 2021 Feb;32(2):218-228. doi: 10.1016/j.annonc.2020.10.600. Epub 2020 Nov 11. PMID 33188874
- [Background] Zhang P, Tong Z, Tian F, Wang Y, Yang J, Li W, Di L, Liu W, Tang L, Qiu R, Xu B. Phase II trial of utidelone as monotherapy or in combination with capecitabine in heavily pretreated metastatic breast cancer patients. J Hematol Oncol. 2016 Aug 11;9(1):68. doi: 10.1186/s13045-016-0297-7. PMID 27516093
- [Background] Zhang P, Sun M, Qiu R, Tang L, Dou G, Xu B. Phase I clinical and pharmacokinetic study of UTD1, a genetically engineered epothilone analog in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2011 Oct;68(4):971-8. doi: 10.1007/s00280-011-1571-6. Epub 2011 Feb 9. PMID 21305287
- [Background] Bollag DM, McQueney PA, Zhu J, Hensens O, Koupal L, Liesch J, Goetz M, Lazarides E, Woods CM. Epothilones, a new class of microtubule-stabilizing agents with a taxol-like mechanism of action. Cancer Res. 1995 Jun 1;55(11):2325-33. PMID 7757983
- [Background] Gerth K, Bedorf N, Hofle G, Irschik H, Reichenbach H. Epothilons A and B: antifungal and cytotoxic compounds from Sorangium cellulosum (Myxobacteria). Production, physico-chemical and biological properties. J Antibiot (Tokyo). 1996 Jun;49(6):560-3. doi: 10.7164/antibiotics.49.560. PMID 8698639
- [Background] Hirte H, Kennedy EB, Elit L, Fung Kee Fung M. Systemic therapy for recurrent, persistent, or metastatic cervical cancer: a clinical practice guideline. Curr Oncol. 2015 Jun;22(3):211-9. doi: 10.3747/co.22.2447. PMID 26089720
- [Background] 2021 ESMO 782P - A retrospective study of toripalimab combined with concurrent chemoradiotherapy in patients with recurrent/advanced cervical cancer.Annals of Oncology (2021) 32 (suppl_5): S725-S772. 10.1016/annonc/annonc703.
- [Background] Peng Peng，Hairong Yao，Dantong Liu，et al.Toripalimab combined with bevacizumab and chemotherapy for refractory, recurrent or metastatic cervical cancer: preliminary results of a single-arm, open-label, phaseⅡtrial. 2023 SGO Annual Meeting on Women's Cancer Abstracts, LBA.
- [Background] Wei XL, Ren C, Wang FH, Zhang Y, Zhao HY, Zou BY, Wang ZQ, Qiu MZ, Zhang DS, Luo HY, Wang F, Yao S, Xu RH. A phase I study of toripalimab, an anti-PD-1 antibody, in patients with refractory malignant solid tumors. Cancer Commun (Lond). 2020 Aug;40(8):345-354. doi: 10.1002/cac2.12068. Epub 2020 Jun 26. PMID 32589350
- [Background] Tang B, Chi Z, Guo J. Toripalimab for the treatment of melanoma. Expert Opin Biol Ther. 2020 Aug;20(8):863-869. doi: 10.1080/14712598.2020.1762561. Epub 2020 May 14. PMID 32406293
- [Background] Alberts DS, Blessing JA, Landrum LM, Warshal DP, Martin LP, Rose SL, Bonebrake AJ, Ramondetta LM. Phase II trial of nab-paclitaxel in the treatment of recurrent or persistent advanced cervix cancer: A gynecologic oncology group study. Gynecol Oncol. 2012 Dec;127(3):451-5. doi: 10.1016/j.ygyno.2012.09.008. Epub 2012 Sep 14. PMID 22986144
- [Background] An J, Li X, Wang J, Zhu L, An R, Jiang K, Huang Y, Wang K, Li G, Wang C, Yuan J, Hou X, Yang G, Li J, Wang Q, Zhu J, Wu L. Efficacy and safety of serplulimab plus nab-paclitaxel in previously treated patients with PD-L1-positive advanced cervical cancer: a phase II, single-arm study. Front Immunol. 2023 Apr 21;14:1142256. doi: 10.3389/fimmu.2023.1142256. eCollection 2023. PMID 37153587
- [Background] Tewari KS, Monk BJ, Vergote I, Miller A, de Melo AC, Kim HS, Kim YM, Lisyanskaya A, Samouelian V, Lorusso D, Damian F, Chang CL, Gotovkin EA, Takahashi S, Ramone D, Pikiel J, Mackowiak-Matejczyk B, Guerra Alia EM, Colombo N, Makarova Y, Rischin D, Lheureux S, Hasegawa K, Fujiwara K, Li J, Jamil S, Jankovic V, Chen CI, Seebach F, Weinreich DM, Yancopoulos GD, Lowy I, Mathias M, Fury MG, Oaknin A; Investigators for GOG Protocol 3016 and ENGOT Protocol En-Cx9. Survival with Cemiplimab in Recurrent Cervical Cancer. N Engl J Med. 2022 Feb 10;386(6):544-555. doi: 10.1056/NEJMoa2112187. PMID 35139273
- [Background] Oaknin A, Gladieff L, Martinez-Garcia J, Villacampa G, Takekuma M, De Giorgi U, Lindemann K, Woelber L, Colombo N, Duska L, Leary A, Godoy-Ortiz A, Nishio S, Angelergues A, Rubio MJ, Farinas-Madrid L, Yamaguchi S, Lorusso D, Ray-Coquard I, Manso L, Joly F, Alarcon J, Follana P, Romero I, Lebreton C, Perez-Fidalgo JA, Yunokawa M, Dahlstrand H, D'Hondt V, Randall LM; ENGOT-Cx10-GEICO 68-C-JGOG1084-GOG-3030 Investigators. Atezolizumab plus bevacizumab and chemotherapy for metastatic, persistent, or recurrent cervical cancer (BEATcc): a randomised, open-label, phase 3 trial. Lancet. 2024 Jan 6;403(10421):31-43. doi: 10.1016/S0140-6736(23)02405-4. Epub 2023 Dec 1. PMID 38048793
- [Background] Colombo N, Dubot C, Lorusso D, Caceres MV, Hasegawa K, Shapira-Frommer R, Tewari KS, Salman P, Hoyos Usta E, Yanez E, Gumus M, Olivera Hurtado de Mendoza M, Samouelian V, Castonguay V, Arkhipov A, Toker S, Li K, Keefe SM, Monk BJ; KEYNOTE-826 Investigators. Pembrolizumab for Persistent, Recurrent, or Metastatic Cervical Cancer. N Engl J Med. 2021 Nov 11;385(20):1856-1867. doi: 10.1056/NEJMoa2112435. Epub 2021 Sep 18. PMID 34534429
- [Background] Colombo N et al. Pembrolizumab plus chemotherapy versus placebo plus chemotherapy for persistent, recurrent, or metastatic cervical cancer: randomized, double-blind, phase 3 KEYNOTE-826 study. ESMO Congress 2021, Abstract LBA2.
- [Background] Monk BJ, Sill MW, McMeekin DS, Cohn DE, Ramondetta LM, Boardman CH, Benda J, Cella D. Phase III trial of four cisplatin-containing doublet combinations in stage IVB, recurrent, or persistent cervical carcinoma: a Gynecologic Oncology Group study. J Clin Oncol. 2009 Oct 1;27(28):4649-55. doi: 10.1200/JCO.2009.21.8909. Epub 2009 Aug 31. PMID 19720909
- [Background] Tewari KS, Monk BJ. Gynecologic oncology group trials of chemotherapy for metastatic and recurrent cervical cancer. Curr Oncol Rep. 2005 Nov;7(6):419-34. doi: 10.1007/s11912-005-0007-z. PMID 16221379
- [Background] Monk BJ, Tewari KS. Invasive cervical cancer. In: DiSaia PJ, Creasman WT, editors. Clinical Gynecologic Oncology. ed 7. Philadelphia, PA: Mosby; 2007. pp. 55-124.
- [Background] Cancer Stat Facts: Cervical Cancer. Available at: https://seer.cancer.gov/statfacts/html/cervix.html. Accessed July 3, 2024.
- [Background] Gennigens C, Jerusalem G, Lapaille L, De Cuypere M, Streel S, Kridelka F, Ray-Coquard I. Recurrent or primary metastatic cervical cancer: current and future treatments. ESMO Open. 2022 Oct;7(5):100579. doi: 10.1016/j.esmoop.2022.100579. Epub 2022 Sep 13. PMID 36108558
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- See also: Cancer Stat Facts: Cervical Cancer — https://seer.cancer.gov/statfacts/html/cervix.html